CLINICAL TRIAL: NCT03922620
Title: Liposomal Bupivacaine vs Peripheral Nerve Block
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Additional published information on the topic since starting the study
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0486
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Results first posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-01

CONDITIONS: Pain, Acute; Surgery; Anesthesia; Opioid Use
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal Bupivacaine Group (Experimental): No peripheral nerve block will be given. Local infiltration of 20cc of Liposomal Bupivacaine infiltrated to the surgical area.
  Interventions: Drug: Liposomal bupivacaine
- Peripheral Nerve Block Group (Active Comparator): Peripheral Nerve Block performed by anesthesia team (blocks will be given by same anesthesia provider utilizing same technique every time in order to reduce variations in delivery of peripheral nerve block). No local analgesic agent infiltration
  Interventions: Drug: Peripheral Nerve Block

INTERVENTIONS:
Drug: Liposomal bupivacaine — Local infiltration of 20cc of Liposomal Bupivacaine infiltrated to the surgical area
  Arms: Liposomal Bupivacaine Group
Drug: Peripheral Nerve Block — Peripheral Nerve Block performed by anesthesia team (blocks will be given by same anesthesia provider utilizing same technique every time in order to reduce variations in delivery of peripheral nerve block).
  Arms: Peripheral Nerve Block Group

SUMMARY:
Liposomal bupivacaine has gained interest in recent literature for its potential to be an effective adjunct to other pain control modalities in a multi-modal approach to post-operative pain control. The goal of this investigation is to compare the efficacy of local administration of liposomal bupivacaine versus the efficacy of a peripheral nerve block in terms of post-operative pain scores after elective ankle and hindfoot surgery. The investigators hypothesize that there will not be a significant difference in the pain scores of these two groups in opioid naïve patients.

DETAILED DESCRIPTION:
Liposomal bupivacaine has gained interest in recent literature for its potential to be an effective adjunct to other pain control modalities in a multi-modal approach to post-operative pain control. Liposomal bupivacaine is an analgesic that is suspended in lipids to allow for gradual release of the analgesic over a 72-hour period (NAMDARI). From prior literature, the utilization of local analgesics infiltrated into surgical sites have been shown to reduce pain in the immediate post-operative period in foot and ankle surgery (GADEK). However, the evaluation of liposomal bupivacaine in foot and ankle surgery is limited. One prospective study found that the addition to liposomal bupivacaine to a multi-modal pain management protocol for forefoot surgery resulted in decreased pain scores during the first four post-operative days as well as fewer refills of opioid pain medication prescriptions, although both findings were not statically significant (ROBBINS). As the general medical community and public policy makers continue to focus on decreasing the amount of opioid pain medications prescribed and available in the community due to the opioid epidemic, liposomal bupivacaine has the potential to be a useful adjunct in the management of post-operative pain without reliance on opioid prescriptions. The goal of this investigation is to compare the efficacy of local administration of liposomal bupivacaine versus the efficacy of a peripheral nerve block in terms of post-operative pain scores after elective ankle and hindfoot surgery. The investigators hypothesize that there will not be a significant difference in the pain scores of these two groups in opioid naïve patients. Furthermore, this study aims to determine if there are differences in the amount of opioid medications utilized for post-operative pain control, patient satisfaction scores, functional outcomes, complications, and unscheduled healthcare contact between the two groups. In order to accomplish these aims, a randomized, controlled investigation will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. Patients undergoing elective primary ankle or hindfoot surgery (ankle arthrodesis, subtalar arthrodesis, triple arthrodesis, total ankle arthroplasty, peroneal tendon debridement/transfer, Cavus Reconstruction, Medial Displacement Calcaneal Osteotomy, Dwyer Osteotomy)

Exclusion Criteria:

1. Patients who are undergoing revision surgical procedure
2. Patients who have taken opioid pain medications in the past 3 months prior to surgical procedure
3. Patients who have allergies to any of the medications or components of medications investigated in the study
4. Patients currently incarcerated
5. Patients who cannot read and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Cush, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Woodbine, Danville, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine Group | Peripheral Nerve Block Group
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Data and outcome measures not tabulated due to discontinued enrollment. | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 baseline participant included as only 1 total participant was enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine Group | Peripheral Nerve Block Group | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (0) |  | 48 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Pain Score
Description: Best 0-10 worst - Continuous scale to measure current pain level
Time Frame: Baseline and 6 weeks
Population: One participant analyzed at baseline as only one total participant was enrolled. No data was displayed at 6 weeks time frame because data was not collected by investigator(s)."
Measure: Number; unit: score on a scale
Arm/Group | Liposomal Bupivacaine Group | Peripheral Nerve Block Group
Number analyzed (Participants) | 1 | 0
score on a scale
  Baseline | 6 |
  6 weeks: number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Morphine Equivalents
Description: morphine equivalents consumed for post-operative pain control
Time Frame: 0-6 weeks
Population: Data was not collected by investigator(s).
Arm/Group | Liposomal Bupivacaine Group | Peripheral Nerve Block Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Investigator-developed, Pain Satisfaction Score
Description: asks patients to rate their level of satisfaction with their pain control on a scale of 0-10, 0 being not satisfied at all and 10 being highly satisfied
Time Frame: 0-6 weeks
Population: Data was not collected by investigator(s).
Arm/Group | Liposomal Bupivacaine Group | Peripheral Nerve Block Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Range of Motion
Description: range of motion measured using goniometer
Time Frame: 0-6 weeks
Population: Data was not collected by investigator(s).
Arm/Group | Liposomal Bupivacaine Group | Peripheral Nerve Block Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Complications
Description: complications after surgery including infection and delayed healing
Time Frame: 6 weeks
Population: One participant analyzed as only one total participant was enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine Group | Peripheral Nerve Block Group
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Unscheduled Healthcare Contact
Description: unscheduled healthcare contact includes patient calls/messages, emergency room visits, or scheduled clinic visits
Time Frame: 6 weeks
Population: One participant analyzed as only one total participant was enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine Group | Peripheral Nerve Block Group
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of surgery to 6-weeks post surgery.
Description: An adverse event (AE) is any untoward, undesired, or unplanned event in the form of signs, symptoms, disease, or laboratory or physiologic observations occurring in a person given a test article or in a clinical study. The event does not need to be causally related to the test article or clinical study.
Arm/Group | Liposomal Bupivacaine Group | Peripheral Nerve Block Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT03922620/Prot_001.pdf